CLINICAL TRIAL: NCT02822430
Title: Pain in Psychiatry : Impact on Length of Hospital Stays
Acronym: D-PSY
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31-13-7017
Record Dates: First submitted 2016-06-21; First posted 2016-07-04 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-06

CONDITIONS: Pain
Keywords: Pain; Psychiatric disorders
MeSH Terms: conditions — Pain; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: Patients with psychiatric disorders will be assessed using five evaluation of pain scales :
  * Visual analogic scale pain
  * Pain behaviour scale
  * Short-FormHealth Survey (SF-36)
  * Global Clinical Impression (GCI) for severity and improvement
  * Mini International Neuropsychiatric Interview (MINI)
  Interventions: Other: Pain scales

INTERVENTIONS:
Other: Pain scales — * Visual analogic scale of pain
  * Pain behaviour scale
  * Short-FormHealth Survey (SF-36)
  * Clinical Global impression
  * Mini International Neuropsychiatric Interview (MINI)

SUMMARY:
For several decades, authors are interested in the existence and meaning of painful symptoms in a population of psychiatric inpatients. But, to date, studies specifically focused on the impact of pain in patient populations in psychiatric hospitals are few. More recently, a review of the literature highlights the difficulties of evaluation of pain in populations of psychiatric patients but also the complex interrelationships between painful symptoms and psychiatric diseases. The first national survey conducted among 172 health which evaluate pain and its management in the field of psychiatry concluded on the need to develop research in this area.

DETAILED DESCRIPTION:
Pain in all the populations remains a major public health issue. Patients with mental illness consult less their general practitioners while they have an increased risk of physical disease. In addition, they have a net reduction in life expectancy due to their mental illness, living conditions and drug treatments.

In this particular population, doctors faces especially difficulties assessment and treatment of pain. Indeed, there is for example in some of these patients difficulties to express that pain.

These painful events make more complex the care of hospitalized patients (eg interrelationship between pain complaints and psychiatric symptoms) and seem to lengthen their hospital stay. This is not without consequences as long as hospitalizations represent an obstacle to the patients psychosocial rehabilitation (installation of daytime activities, project work rehabilitation, development of social network ...) and impair their quality of life.

And for the patients with psychiatric disorders some points can be noticed :

* An increased risk of physical disease
* Warning signs like pain poorly known and poorly evaluated ... and poorly supported
* The presence of the pain seems to lengthen the hospital stay
* An extension of the hospital stay, which represent an obstacle to the psychosocial rehabilitation This research project is to test if the presence of a painful complaint among psychiatric inpatients is associated lengthening of the hospitalization duration.

The secondary objectives of this study are:

* To measure the prevalence of painful complaint in this specific population,
* To examine the evolution of pain during hospitalization.
* Identify factors influencing the relationship between pain and length of stay
* To identify if the intensity of the psychiatric illness is associated with pain intensity measured

Confirmation of these objectives would lead to a better understanding of the factors influencing psychiatric hospital stays and thus more efficient management of health resources.

In addition, the present study will well identify and implement standardized assessments of pain for these patients.

For these patients the interest is important because they can be in great difficulty to express a painful complaint. These people have often difficulties to communicate, and live in a sometimes precarious environment and severity of disorders reduce their access to care.

This approach is part of a comprehensive approach taking account of the psychiatric and somatic disorders in a very vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Patient eighteen years old
* Patient hospitalized in psychiatric service at Toulouse University Hospital
* Informed consent signed

Exclusion Criteria:

* Patient treated with maintenance sismotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with psychiatric disorders
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2014-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Influence of pain on hospitalization stay evaluated with pain visual analogic scale | Day 1
  Multivariate regression analysis
Influence of pain on hospitalization stay evaluated with pain visual analogic scale | Day 7
  Multivariate regression analysis
Influence of pain on hospitalization stay evaluated with pain visual analogic scale | 2 days before patient end of hospitalization
  Multivariate regression analysis

SECONDARY OUTCOMES:
Evaluation of pain in psychiatric population with visual analogic scale of pain | Day 1
Evaluation of pain in psychiatric population with visual analogic scale of pain | Day 7
Evaluation of pain in psychiatric population with visual analogic scale of pain | 2 days before patient end of hospitalization
Evaluation of pain intensity impact on Mini International Neuropsychiatric Interview score | Day 1
Evaluation of pain intensity impact on Mini International Neuropsychiatric Interview score | 2 days before the patient end of hospitalization
Evaluation of gender impact on pain intensity using visual analogic scale of pain | Day 1
Evaluation of gender impact on pain intensity using visual analogic scale of pain | 2 days before the patient end of hospitalization
Evaluation of age impact on pain intensity using visual analogic scale of pain | Day 1
Evaluation of age impact on pain intensity using visual analogic scale of pain | 2 days before the patient end of hospitalization
Evaluation of Mini International Neuropsychiatric Interview score impact on hospitalization stay | Day 1
Evaluation of Mini International Neuropsychiatric Interview score impact on hospitalization stay | 2 days before the patient end of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Laurent SCHMITT, PHD, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Functionnal unit of psychiatry, Toulouse, France

IPD SHARING:
Plan to Share IPD: No